CLINICAL TRIAL: NCT06098157
Title: Tuebingen Register of Union Failure After Fractures of the Upper and Lower Extremities
Acronym: TRUFFLE
Status: Recruiting | Type: Observational
Sponsor: Department of Trauma and Reconstructive Surgery at Eberhard Karls University Tuebingen, BG Klinik Tu (Other)
Responsible Party: Principal Investigator, Marie K. Reumann, Principal Investigator, Head of Clinical Trauma Research, Department of Trauma and Reconstructive Surgery at Eberhard Karls University Tuebingen, BG Klinik Tu
Other Study IDs: TRUFFLE
Record Dates: First submitted 2023-09-28; First posted 2023-10-24 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-11

CONDITIONS: Pseudarthrosis; Ununited Fracture
Keywords: bone; non-union; delayed union; delayed bone healing; pseudarthrosis; callus formation; ununited fracture; fracture healing
MeSH Terms: conditions — Pseudarthrosis; Fractures, Ununited

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
TRUFFLE is a register of clinical patient data of failed bone healing and bone non-union after fracture. All patients suffering from a long bone delayed or non-union after fracture and undergoing revision surgery are registered with their clinical data, comorbidities, medication, soft tissue status, radiographic status, Non-Union Scoring System (NUSS) Score and are followed up until final bone healing or end of treatment. The register consists of more than 800 patients cases. The aim is to identify risk factors for healing of non-unions. Data analysis will compare those patients that undergo regular healing to those of insufficient healing.

DETAILED DESCRIPTION:
Bone non-union is a severe complication in trauma surgery. It requires complex surgical intervention leading to decisive restrictions for the patient as well as socioeconomic burden for the health care systems. Despite extensive research, up to date, bone healing has not yet been fully understood. Many risk factors impairing bone healing causing delayed healing or even non-union after fracture have been studied in the past. However, these studies mainly focus on secondary and tertiary prevention measures id est when fracture healing is delayed or the non-union is already present. Research concerning the identification of risk factors concerning primary prevention of non-healing after non-union treatment are scarce, usually investigate a certain anatomical location. Also, as the incidence of non-union (5 % to 10 %) is very low, these studies often only include a limited number of cases and brief follow-up periods.

Thus, TRUFFLE was started as a register for non-union cases aiming for large number of patients cases with consisted data and a follow-up period till the end of treatment.

All patients suffering from a long bone delayed or non-union after fracture and undergoing revision surgery are registered with their clinical data, comorbidities, medication, soft tissue status, radiographic status, Non-Union Scoring System (NUSS) Score and are followed up until final bone healing or end of treatment. The register consists of more than 800 patients cases.

All parameters examined are evaluated at the time of non-union index procedure. Data include demographic parameters as age and gender, type of primary injury according to classification of the AO foundation, severity of primary injury (injury severity score (ISS) > 16), Gustilo-Anderson classification at the time of initial trauma, presence of traumatic brain injury, number of previous soft tissue surgeries before non-union index procedure. The state of infection of the designated bone segment stated by proof of microbiological colonization at the time of non-union index procedure is assessed, as well as Weber/Cech classification of non-union. Comorbidities such as diabetes mellitus, cardiovascular disease, rheumatological conditions, cancer and neurological disease (i.e. Parkinson's disease), as well as tobacco smoking and classification according to the American Society of Anesthesiologists (ASA classification) are assessed. Intake of medication and lab parameters are listed. Any subsequent revision surgery related to the designated non-union is included during patients follow-up. The NUSS- Score is evaluated and calculated according to above listed parameters. Also, subjective parameters of patients quality of life are included at non-union index procedure and at subsequent follow-ups.

Bone healing or unsuccessful healing serve as primary outcome parameter as well as time to heal.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* presence of long bone non-union that required surgical treatment.
* radiological signs according to the criteria of the Radiographic Union Scale of Tibial fractures (RUST).
* clinical signs as pain, lack of weight bearing and/or limitation on range of motion.

Exclusion Criteria:

* age <18 years
* Patients with non surgical intervention and presence of long bone non-union
* bone non-union that resulted from elective orthopedic surgery (e.g. osteotomies).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for delayed bone healing or non-union in a level 1 hospital of maximum trauma care
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
number of participants with successful bone healing | minimum of 1 year up to 5 years after non-union index procedure
  End of treatment can either be successful healing or treatment with no success in bone healing (i.e. amputation, total joint replacement). The number of participants reaching successful healing (responders) to those who are not reaching successful healing (non-responders) will be analyzed.
Time to heal | minimum of 1 year up to 5 years after non-union index procedure
  Time to heal is defined as the length of time from non-union index procedure to date of last follow-up visit that stated radiographic and clinical success or unsuccessful bone healing (i.e. amputation, total joint replacement).

SECONDARY OUTCOMES:
Charlson Comorbidity Index | minimum of 1 year up to 5 years after non-union index procedure
  Comorbidities are listed according to the Charlson Comorbidity Index, at time of non-union index procedure. 19 comorbidities and patients age are listed according to which a score from 0 to > 5 is calculated. A 1 - year mortality risk is predicted. The higher the score from 0 to 5 combined with increasing age, the higher the risk of mortality, with 0 as the lowest score with the lowest risk, and > 5 as the highest score with the highest risk.
number of medication | minimum of 1 year up to 5 years after non-union index procedure
  any intake of medication at time of non-union index procedure is listed. The number of medications are evaluated.
number of participants undergoing type of revision surgery | minimum of 1 year up to 5 years after non-union index procedure
  number of participants undergoing several types of revision surgery (plate, nail, external fixation, autologous bone grafting) at time of non-union index procedure
number of participants suffering from local infection | minimum of 1 year up to 5 years after non-union index procedure
  number of participants suffering from type of local infection at time of non-union index procedure is listed. Microbiological tests can reveal bacterial infection. Any sort of bacterial infection of local soft tissue and bone non-union according to microbiological tests are listed and qualify for infection (yes or no).
NUSS - non union scoring system | minimum of 1 year up to 5 years after non-union index procedure
  All individual parameters of the 3 categories within the NUSS (bone-, patient- soft tissue related) are captured. A maximum score of 100 points can be scored. The score is related to 4 risk groups according to the number of points reached. The higher the number the points the higher is the risk group (1 - 25 points for risk group 1, 26 - 50 points for risk group 2, 51 - 75 points for risk group 3, 76 - 100 points for risk group 4). A surgical procedure is suggested according to the risk group with only limited surgical intervention in risk group 1 and increasing invasiveness for risk groups with higher scores (2, 3 and 4). Risk group 4 with the highest score level suggest severe surgical interventions (i.e. amputation or total joint implantation).
  The NUSS and subsequent risk group - levels are analyzed at time of non-union index procedure and any subsequent follow up visit that requires a surgical procedure.
Weber Cech classification | minimum of 1 year up to 5 years after non-union index procedure
  Weber Cech classification (atrophic, hypertrophic, oligotrophic) at time of non-union index procedure
patient reported outcome measures (PROMS) | minimum of 1 year up to 5 years after non-union index procedure
  The EQ5D5L, a standardized measure of health-related quality of life developed by the EuroQol Group with 5 dimensions and 5 levels, is assessed by the patient at time of non-union index procedure and every follow- up visit. A score from 1 to 5 can be reached with 1 being the lowest, and 5 being the highest score. The higher the score the worse is the health state of the participant.
ASA (American Society of Anesthesiologists) classification | minimum of 1 year up to 5 years after non-union index procedure
  The ASA Score (I - VI) measures the physical status of a patients before surgical intervention.
  ASA I represents a good state of health, while ASA VI represents a very severe state of health (i.e. a declared brain dead person). It is assessed at time of non-union index procedure and before any subsequent follow- up surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Marie K Reumann, MD, Study Director — Department of Trauma and Reconstructive Surgery at Eberhard Karls University Tuebingen
Locations (1):
- Department of Trauma and Reconstructive Surgery at Eberhard Karls University Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No